CLINICAL TRIAL: NCT02777372
Title: Psychophysiology, Neurosteroids, and Stress in Premenstrual Dysphoric Disorder
Brief Title: Stress & Premenstrual Symptoms Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00220794; 1K23MH107831-01A1 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-05-19 (Estimated); Results first posted 2022-11-17 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: PMDD; Stress; Mood
Keywords: Zoloft; premenstrual syndrome (PMS); Menses
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline (Experimental): To determine the impact of short term luteal phase treatment with Sertraline 50mg tablets (PMDD group only) on acoustic startle response across the menstrual cycle. Sertraline 50 mg tablets are administered daily from ovulation until menses onset.
  Interventions: Drug: Sertraline
- Control (No Intervention): No intervention.

INTERVENTIONS:
Drug: Sertraline — Sertraline will be provided at a dose of 50 mg daily for up to 3 weeks, depending on the length of a woman's luteal phase. Medication will be taken only during the luteal phase. Women will initiate sertraline treatment upon determining that they have ovulated (using a urine luteinizing hormone (LH) Kit) and remain on sertraline until onset of their next menstrual period at which time they will stop taking the medication.
  Other Names: Zoloft
  Arms: Sertraline

SUMMARY:
This study that aims to evaluate the psychophysiology of premenstrual mood disorders (PMDs) at baseline and after treatment with sertraline. Participants will include women with PMDs and healthy female controls. Participation involves a baseline visit to determine eligibility and three study visits that include questionnaires and stress reactivity assessment via an acoustic startle paradigm. Female participants with PMDs will receive sertraline during the premenstrual phase.

DETAILED DESCRIPTION:
Among women with premenstrual mood dysphoric disorder (PMDD), baseline arousal is heightened during the luteal phase of the menstrual cycle compared to the follicular phase, as measured by acoustic startle response (ASR). Healthy female controls do not show cyclic changes in this measure of physiologic arousal. It has been suggested that such heightened physiologic arousal during the luteal phase may be due to differences in neurosteroid modulation of Gamma-aminobutyric acid (GABA)-A receptor function. Research indicates that women with premenstrual mood disorders (PMDs) may have sub-optimal sensitivity to the progesterone metabolite allopregnanolone (ALLO), a GABA-A receptor modulator. In animal models, intracerebroventricular injection of corticotrophin releasing factor (CRF) increases amplitude of the acoustic startle response, while ALLO administration attenuates this CRF-enhanced startle. The primary aim of this study is to examine differences in ASR by menstrual cycle phase (follicular, luteal) and group (control, PMDD). Secondary aim is to examine the impact of luteal phase treatment with a selective serotonin reuptake inhibitor (SSRI) on psychophysiology in women with PMDs. An exploratory aim is to examine immune function among these women.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

1. Aged 18 - 50 years, per self-report
2. Able to give written informed consent, per self-report
3. Fluent in written and spoken English
4. Have normal or corrected to normal hearing and vision, per self-report
5. Female participants must be experiencing regular menstrual cycles (24-39 days), per self-report
6. Have a negative urine drug screen.

Exclusion Criteria:

Participants cannot have:

1. Use of an psychotropic medication anytime in the past 2 months, per self-report
2. Drug or alcohol abuse history within previous 2 years
3. Lifetime history of psychotic disorder including, schizophrenia, schizoaffective disorder, major depression with psychotic features and bipolar disorder, per self-report
4. Currently homeless, per self-report
5. History of any Axis I disorder other then specific phobia within the past 12 months, per Structured Clinical Interview for Diagnostic and Statistical Manual (SCID) interview
6. Active suicidal ideation (suicide plan or suicide attempt) within the previous 6 months, per self-report
7. Steroid hormone or hormonal contraceptive use in the past 6 months, per self-report, except emergency contraceptive use
8. Pregnancy in the past year, per self-report. Pregnancy during the study is also exclusionary. Participants must use a reliable, nonhormonal form of birth control during the study. If a participant becomes pregnant, she must inform study staff.
9. Sensitive hearing, per self-report.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Hantsoo, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Center for Women's Reproductive Mental Health, Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epperson CN, Pittman B, Czarkowski KA, Stiklus S, Krystal JH, Grillon C. Luteal-phase accentuation of acoustic startle response in women with premenstrual dysphoric disorder. Neuropsychopharmacology. 2007 Oct;32(10):2190-8. doi: 10.1038/sj.npp.1301351. Epub 2007 Feb 21. PMID 17314917
- [Background] Hantsoo L, Epperson CN. Premenstrual Dysphoric Disorder: Epidemiology and Treatment. Curr Psychiatry Rep. 2015 Nov;17(11):87. doi: 10.1007/s11920-015-0628-3. PMID 26377947
- [Background] Epperson CN, Hantsoo LV. Making Strides to Simplify Diagnosis of Premenstrual Dysphoric Disorder. Am J Psychiatry. 2017 Jan 1;174(1):6-7. doi: 10.1176/appi.ajp.2016.16101144. No abstract available. PMID 28041003
- [Background] Hantsoo L, Golden CEM, Kornfield S, Grillon C, Epperson CN. Startling Differences: Using the Acoustic Startle Response to Study Sex Differences and Neurosteroids in Affective Disorders. Curr Psychiatry Rep. 2018 May 18;20(6):40. doi: 10.1007/s11920-018-0906-y. PMID 29777410
- [Background] Hantsoo L, Epperson CN. Allopregnanolone in premenstrual dysphoric disorder (PMDD): Evidence for dysregulated sensitivity to GABA-A receptor modulating neuroactive steroids across the menstrual cycle. Neurobiol Stress. 2020 Feb 4;12:100213. doi: 10.1016/j.ynstr.2020.100213. eCollection 2020 May. PMID 32435664
- [Result] Hantsoo, L., Kaminsky, Z., Payne, J.L. Luteal Phase Epigenetic Biomarkers Identify Premenstrual Dysphoric Disorder (PMDD) and Selective Serotonin Reuptake Inhibitor (SSRI) Response in PMDD. Neuropsychopharmacology (2022) 47:220 - 370.
- [Result] Miller KN, Standeven L, Morrow AL, Payne JL, Epperson CN, Hantsoo L. GABAergic neuroactive steroid response to sertraline in premenstrual dysphoric disorder. Psychoneuroendocrinology. 2024 Feb;160:106684. doi: 10.1016/j.psyneuen.2023.106684. Epub 2023 Nov 30. PMID 38091917
- [Result] Barone JC, Ho A, Osborne LM, Eisenlohr-Moul TA, Morrow AL, Payne JL, Epperson CN, Hantsoo L. Luteal phase sertraline treatment of premenstrual dysphoric disorder (PMDD): Effects on markers of hypothalamic pituitary adrenal (HPA) axis activation and inflammation. Psychoneuroendocrinology. 2024 Nov;169:107145. doi: 10.1016/j.psyneuen.2024.107145. Epub 2024 Jul 24. PMID 39096755
- [Result] Hantsoo L, Grillon C, Sammel M, Johnson R, Marks J, Epperson CN. Response to sertraline is associated with reduction in anxiety-potentiated startle in premenstrual dysphoric disorder. Psychopharmacology (Berl). 2021 Oct;238(10):2985-2997. doi: 10.1007/s00213-021-05916-6. Epub 2021 Jul 22. PMID 34292344

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Controls do not receive sertraline.
- Sertraline: To determine the impact of short term luteal phase treatment with Sertraline 50mg tablets (PMD group only) on arousal regulation across the menstrual cycle.
  Sertraline: Sertraline will be provided at a dose of 50 mg daily for up to 3 weeks, depending on the length of a woman's luteal phase. Medication will be taken only during the luteal phase. Women will initiate sertraline treatment upon determining that they have ovulated (using a urine luteinizing hormone (LH) Kit) and remain on sertraline until onset of their next menstrual period at which time they will stop taking the medication.
Period: Overall Study
Arm/Group | Control | Sertraline
Started | 43 | 41
Completed | 24 | 23
Not Completed | 19 | 18

BASELINE CHARACTERISTICS:
Groups:
- Sertraline: To determine the impact of short term luteal phase treatment with Sertraline 50mg tablets (PMD group only) on arousal regulation across the menstrual cycle.
  Sertraline: Sertraline will be provided at a dose of 50 mg daily for up to 3 weeks, depending on the length of a woman's luteal phase. Medication will be taken only during the luteal phase. Women will initiate sertraline treatment upon determining that they have ovulated (using a urine LH Kit) and remain on sertraline until onset of their next menstrual period at which time they will stop taking the medication.
- Total: Total of all reporting groups
Arm/Group | Control | Sertraline | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 41 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (6.3) | 33.6 (7.7) | 30.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 41 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 20 | 23 | 43
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 41 | 84

OUTCOME MEASURES:

1. Primary Outcome: Acoustic Startle Response (ASR) Magnitude Based on Menstrual Cycle Phase
Description: Acoustic startle response (ASR) is measured during the follicular and luteal phase of the menstrual cycle in controls and those with PMDD. Magnitude of ASR is measured using the eyeblink reflex, by recording activity from the orbicularis oculi muscle. Recording is performed via two surface disk electrodes (Ag-AgCl) applied underneath the left eye; one in line with the pupil and one 1-2 cm lateral to the first one. For the primary outcome of baseline ASR magnitude over the menstrual cycle, peak amplitude of the blink reflex was determined in the 20-120-ms time frame following stimulus onset relative to baseline (baseline is the average baseline electromyography (EMG) level for the 50 ms immediately preceding auditory stimulus onset). ASR is measured in microvolts, and raw ASR results are standardized to t-scores. Higher ASR t-score indicates greater contraction of the the orbicularis oculi muscle. A t-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Month 1 (Follicular), Month 2 (Luteal)
Population: 33 Controls and 24 PMDD (Sertraline) completed the Month 1 (Follicular) visit, and 27 Controls and 23 premenstrual mood dysphoric disorder (PMDD) completed the Month 2 (Luteal) visit. Assessments were done on 1 day of the Follicular phase and 1 day of the Luteal phase.
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Control | Sertraline
Number analyzed (Participants) | 33 | 24
t score
  Month 1 (Follicular) | 54.2 (4.4) | 53.7 (4.7)
  Month 2 (Luteal): number analyzed (Participants) | 27 | 23
  Month 2 (Luteal) | 56.4 (4.8) | 53.3 (4.8)
Statistical Analysis 1: Comparison: Control vs Sertraline; Effect of group on differences in ASR t scores from follicular to luteal; Test type: Other; p = 0.139, Regression, Linear

2. Primary Outcome: Impact of Sertraline on ASR Magnitude
Description: This outcome examines the impact of luteal phase treatment with a selective serotonin reuptake inhibitor (SSRI) (PMDD group only) on acoustic startle response (ASR). ASR is measured using the eyeblink reflex, measured by recording activity from the orbicularis oculi muscle. Recording is performed via two surface disk electrodes (Ag-AgCl) applied underneath the left eye; one in line with the pupil and one 1-2 cm lateral to the first one. Peak amplitude of the blink reflex is determined in the 20-120-ms time frame following stimulus onset. PMDD participants complete test day 3 (Luteal Month 3) while on sertraline and their ASR magnitude will be compared to their previous luteal test day (Luteal Month 2). ASR is measured in microvolts, and raw ASR results are standardized to t-scores. Higher ASR t-score indicates greater contraction of the the orbicularis oculi muscle. A t-score of 50 indicates the population mean with a standard deviation of 10.
Time Frame: Month 2 (Luteal), Month 3 (Luteal)
Population: 27 Controls and 23 PMDD (Sertraline) completed Luteal Month 2, and 24 Controls and 23 PMDD completed Luteal Month 3. Assessments were done on 1 day of the Luteal phase in Month 2 and 1 day of the Luteal phase in Month 3.
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | Control | Sertraline
Number analyzed (Participants) | 27 | 23
t score
  Month 2 (Luteal) | 56.4 (4.8) | 53.3 (4.8)
  Month 3 (Luteal): number analyzed (Participants) | 24 | 23
  Month 3 (Luteal) | 51.8 (4.6) | 52.2 (5.0)
Statistical Analysis 1: Comparison: Control vs Sertraline; Test type: Other; p = 0.843, Regression, Linear — Effect of group on ASR t score in the first luteal phase (no medication) to the second luteal phase (sertraline)

3. Secondary Outcome: Interleukin 6 (IL-6) Level
Description: Blood samples were collected to measure serum interleukin-6 (IL-6). IL-6 levels were compared in the follicular and luteal phases, between Control and PMDD groups. Levels are measured in picogram/milliliter (pg/mL).
Time Frame: Month 1 (Follicular ), Month 2 (Luteal )
Population: 38 participants in the Control group and 32 participants in the PMDD group had blood available for IL-6 measurement in the Follicular phase. 36 Controls and 32 PMDD had blood available for IL-6 in the Luteal 1 phase. Assessments were done on 1 day of the Follicular phase and 1 day of the Luteal phase.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Control | Sertraline
Number analyzed (Participants) | 38 | 32
picogram/milliliter (pg/mL)
  Month 1 (Follicular) | 0.4 (0.19) | .34 (.15)
  Month 2 (Luteal): number analyzed (Participants) | 36 | 32
  Month 2 (Luteal) | .59 (.46) | .4 (.17)
Statistical Analysis 1: Comparison: Control vs Sertraline; Test type: Other; p = 0.06, t-test, 2 sided

4. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-alpha) Level
Description: Blood samples were collected to measure serum TNF-alpha levels in the Follicular and Luteal 1 phases. Levels are measured in picogram/milliliter (pg/mL).
Time Frame: Month 1 (Follicular ), Month 2 (Luteal )
Population: 38 Controls and 32 PMDD had blood available to measure TNF-alpha in the Follicular phase. 36 Controls and 32 PMDD had blood available to measure TNF-alpha in the Luteal phase. Assessments were done on 1 day of the Follicular phase and 1 day of the Luteal phase.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Control | Sertraline
Number analyzed (Participants) | 38 | 32
pg/mL
  Month 1 (Follicular ) | 1.27 (.32) | 1.63 (.52)
  Month 2 (Luteal ): number analyzed (Participants) | 36 | 32
  Month 2 (Luteal ) | 1.27 (.36) | 1.54 (.31)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Participants in the control arm were not assessed for adverse events since they did not receive an intervention. Only 23 participants in the sertraline arm stayed on study to be assessed for adverse events.
Groups:
- Sertraline: To determine the impact of short term luteal phase treatment with Sertraline 50mg tablets (PMDD group only) on arousal regulation across the menstrual cycle.
  Sertraline: Sertraline will be provided at a dose of 50 mg daily for up to 3 weeks, depending on the length of a woman's luteal phase. Medication will be taken only during the luteal phase. Women will initiate sertraline treatment upon determining that they have ovulated (using a urine LH Kit) and remain on sertraline until onset of their next menstrual period at which time they will stop taking the medication.
Arm/Group | Control | Sertraline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02777372/Prot_SAP_000.pdf